CLINICAL TRIAL: NCT04035395
Title: Salud y Vida 2.0: Enhancing Integrated Behavioral Health for Individuals With Diabetes in the Rio Grande Valley
Brief Title: Salud y Vida 2.0: Enhancing Integrated Behavioral Health for Diabetics in the Rio Grande Valley
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Health Resources in Action, Inc. (Other)
Responsible Party: Principal Investigator, Belinda Reininger, Professor and Regional Dean, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HSC-SPH-16-0044
Record Dates: First submitted 2019-07-24; First posted 2019-07-29 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-07

CONDITIONS: Diabetes Mellitus, Type 2; Behavior, Health
Keywords: Integrated Behavioral Health; Community Health Workers
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Health Behavior | interventions — Exercise; Nutritional Status

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants were not told whether they had been randomized into the intervention or control group. However, when the participant was offered new intervention services, the participant could infer that they were part of the intervention group. Conversely, if a participant was only offered the standard intervention services, they could infer they were part of the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants randomized to the intervention group will receive the SyV 2.0 program, which in addition to standard diabetes management services of SyV 1.0 services, could include MTM services, care coordination by a team of behavioral health care providers, and/or referrals to community-based lifestyle programs, as determined by their tailored care plan. The participant will be seen by evaluation staff to complete baseline assessment for the study. Then, an individualized care plan will be developed by SyV 1.0 interdisciplinary staff and reviewed by the chronic care case management team. The care plan will include information on additional services provided by UTHealth such as, but not limited to, behavioral health services, or pharmacy services. Each participant will receive an individualized care plan and when applicable, referrals to community-based programs. Evaluation staff and CHWs will make follow-up appointments for the participant depending on their care plan.
  Interventions: Other: Peer-led Support Group; Other: Behavioral Health Consult; Other: Medication Therapy Management Consult; Other: La Cocina Alegre/ The Happy Kitchen; Other: Mind, Exercise, Nutrition, Do it!
- Control (No Intervention): Participants randomized to the usual care group will receive the SyV 1.0 program which includes community based program referrals (excluding intervention programs) and home-based visits from CHWs. These participants will also receive the standard follow-up from UTHealth staff such as a phone call, an information session as per their treatment plan, and /or a onetime mailing of information about the importance of following their treatment plan. Before implementation begins, additional details about standard care will be ascertained from partner organizations to better understand how these differ from the treatment conditions of the intervention group. Once the participant completes 12 months in the study, 2.0 services will be initiated.

INTERVENTIONS:
Other: Peer-led Support Group — The Viviendo Saludable pláticas (or talks) connected Salud y Vida participants living with diabetes together. These talks served as a forum for Salud y Vida participants to share their knowledge and experiences, including some that many health workers, friends, or family do not have. Viviendo Saludable helped participants develop better strategies for managing their diabetes in their daily life. The Viviendo Saludable pláticas complement and enhance the other services by helping participants create a network of emotional, social, and practical support needed to manage diabetes and stay healthy over the long term. Classes met once a week for one hour at locations central to participants' homes.
  Other Names: Viviendo Saludable platicas
  Arms: Intervention
Other: Behavioral Health Consult — In a Behavioral Health consult, a participant meets with a counselor for one or more thorough meetings to talk about things that influence their health and well-being. A participant receiving a Behavioral Health consult receives support and is empowered with health coping skills that will allow for improved medication adherence and motivation to control their diabetes.
  Arms: Intervention
Other: Medication Therapy Management Consult — Medication Therapy Management helps participants and their doctors make sure that their medications are working to improve their health. In a Medication Therapy Management (MTM) consult, a pharmacist gives participants a comprehensive review of all their medications and speaks with them about 1) how well their medications are working, 2) whether their medications have side effects, 3) if there might be interactions between the drugs their taking, 4) whether costs can be lowered and 5) other problems participants are having. The participant will get a written summary of this discussion, including an action plan that recommends what can be done to make the best use of their medications.
  Arms: Intervention
Other: La Cocina Alegre/ The Happy Kitchen — The Happy Kitchen is a program where people come together to learn skills and self-sufficiency in preparing healthy, economical meals, laugh, cook, and enjoy food together. The cooking and nutrition program is an interactive 6-week series of classes, where the essential skills for healthy eating is taught and emphasis is placed on the selection and preparation of fresh, seasonal foods that are nutritious, economical, and delicious. Classes meet once a week for 1 ½ hours to cook, discuss, and learn together. All participants leave each class with recipes and groceries to practice new cooking skills.
  Arms: Intervention
Other: Mind, Exercise, Nutrition, Do it! — MEND is a diet and exercise education program that helps families support their kids, ages 6-13, to reach a healthy weight. The program teaches adults and their children how to maintain energy and confidence throughout the day while learning how to cook healthy meals. Each program lasts 10 weeks and classes are 2 times per week. An adult must attend with the child.
  Arms: Intervention

SUMMARY:
The purpose of this study is to implement a system of integrated health care that provides a continuum of care for those with diabetes. This study will use a randomized behavioral intervention trial experimental design to compare participants receiving the enhanced delivery of integrated behavioral care with nonparticipants receiving the usual care until after the study period, at which time they will be offered access to expansion services.

DETAILED DESCRIPTION:
The Rio Grande Valley (RGV), located on the northern bank of the Rio Grande River that separates the United States from Mexico, is home to more than 1.2 million residents, representing about 5% of Texas' general population. The SyV 2.0 program focuses on the system of health care in the lower RGV, comprised of a predominantly Mexican American, low-income, underserved community with chronic disease rates and related mortality that exceed those in most other regions of the state and the nation. Based on a cohort study of 2,000 Mexican American adults from this region between 2003 to 2008 called the Cameron County Hispanic Cohort (CCHC), researchers estimated diabetes prevalence to be 31% and 81% of the population were either obese (49%) or overweight (32%). Residents in this region suffer from disproportionate health disparities that stem from extreme poverty (40% of families live below federal poverty line), lower levels of educational attainment (9.9 average years of education), and inadequate access to basic health care needs, income, and education.

The SyV 2.0 program is an expansion of SyV 1.0, a program for individuals with uncontrolled diabetes. Enhancement includes two major initiatives: clinical-based services and community-based services. Clinical based services will include medication therapy management for participants with low levels of medication adherence and care coordination which includes behavioral health services for participants who do not qualify for services with the mental health authority, but need behavioral health support. Community-based services will include peer led support groups and access to community-based lifestyle programs (capacity building cooking classes and an obesity awareness program). Clinical-based and community-based services will be directed by a multidisciplinary care team and will be customized to meet each participant's individualized needs.

The proposed study does not pose any major risks or dangers beyond what a normal physician visit would present. Benefits include improved control of chronic disease (diabetes, hypertension, and obesity), a reduction in depression, increased access to behavioral healthcare services, and improved adult functioning and quality of life for current SyV 1.0 participants.

This study will contribute to the investigator's understanding of how to increase access to health care services and treatment among those individuals with diabetes, namely, low-income, Hispanic communities.

* This study was not funded by the National Institutes of Health (NIH). It was funded by two Texas foundations, Methodist Healthcare Ministries and Valley Baptist Legacy Foundation.

ELIGIBILITY:
Inclusion Criteria:

* Participants of the Salud y Vida (SyV) program who are patients at two specific clinics
* Reside in the lower Rio Grande Valley of Texas
* A diagnosis of poorly controlled diabetes (HbA1c greater than or equal to 9.0%)
* Enrollment in the SyV 1.0 services for a minimum of 6 months
* At 6 months still have uncontrolled diabetes (HbA1c greater than or equal to 9.0%)

Exclusion Criteria:

* Enrollment in another research study
* Does not speak either English or Spanish
* Immediate family member of current SyV 2.0 participant
* Not a registered patient at 1 of the 2 specified clinics

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 353 (Actual)
Dates: Start 2016-09-29 (Actual); Primary Completion 2018-06-13 (Actual); Study Completion 2018-06-13 (Actual)

PRIMARY OUTCOMES:
Rate of Change in Hemoglobin A1c | 12 month period
  Participants who receive SyV 2.0 will experience a change in HbA1c after 12 months compared to participants who receive SyV 1.0 (the standard of care).

SECONDARY OUTCOMES:
Rate of Change in Blood Pressure | 12 month period
  Participants who receive SyV 2.0 will experience a change in their blood pressure after 12 months compared to participants who receive SyV 1.0. Both systolic and diastolic pressures will be assessed during the study period.
Rate of Change in BMI | 12 month period
  Participants who receive SyV 2.0 will experience a change in their BMI after 12 months compared to overweight or obese participants who receive SyV 1.0.
Rate of Change in Depressive Symptoms | 12 month period
  Participants who receive SyV 2.0 will experience a change in their depressive symptoms, as measured by the Patient Health Questionnaire-9 (PHQ-9), after 12 months compared to participants who receive SyV 1.0. The PHQ-9 is a multipurpose instrument for screening, diagnosing, monitoring and measuring the severity of depression. The PHQ-9 total possible score is 27. The PHQ-9 scoring criteria is categorized as minimal (0-4), mild (5-9), moderate (10-14), moderately severe (15-19) and severe (20-27) depression. Higher values represent worse outcome.
Rate of Change in Quality of Life: Duke Health Profile | 12 month period
  Participants who receive SyV 2.0 will experience a change in their quality of life, as measured by the Duke Health Profile, after 12 months compared to participants who receive SyV 1.0. The Duke Health Profile is a 17-item generic questionnaire instrument designed to measure adult self-reported functional health status quantitatively during a one-week time window. The Duke Health profile has 11 scales, six of which measure function and five of which measure dysfunction. Scores range from 0 to 100. For scales measuring function, the higher the score, the more functional the person being evaluated. For scales measuring dysfunction, the higher the score, the more dysfunctional the person being evaluated. The general health domain score, a composite of the physical health, mental health and social health domain scores, was utilized as the primary quality of life indicator in our analyses.
Rate of Change in Total Cholesterol | 12 month period
  Participants who receive SyV 2.0 will experience a change in their total cholesterol after 12 months compared to participants who receive SyV 1.0.
Rate of Change in Self-efficacy: Diabetes Self-Efficacy Scale | 12 month period
  Participants who receive SyV 2.0 will experience a change in self-efficacy, as measured by the Diabetes Self-Efficacy Scale, after 12 months compared to participants who receive SyV 1.0. The Diabetes Self-Efficacy Scale is an 8-item generic questionnaire instrument that is self-reported and designed to measure adult patient perception in regard to performing self-care tasks related to diabetes. The Diabetes Self-Efficacy Scale has 8 items. Scores range from 0 to 10. The lower the score, the lower the self-efficacy of the person being evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Belinda M. Reininger, DrPH, Principal Investigator — The University of Texas Health Science Center, Houston

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fisher-Hoch SP, Vatcheva KP, Laing ST, Hossain MM, Rahbar MH, Hanis CL, Brown HS 3rd, Rentfro AR, Reininger BM, McCormick JB. Missed opportunities for diagnosis and treatment of diabetes, hypertension, and hypercholesterolemia in a Mexican American population, Cameron County Hispanic Cohort, 2003-2008. Prev Chronic Dis. 2012;9:110298. doi: 10.5888/pcd9.110298. PMID 22863308
- [Derived] Reininger BM, Lee M, Hessabi M, Mitchell-Bennett LA, Sifuentes MR, Guerra JA, Ayala CD, Xu T, Polletta V, Flynn A, Rahbar MH. Improved diabetes control among low-income Mexican Americans through community-clinical interventions: results of an RCT. BMJ Open Diabetes Res Care. 2020 May;8(1):e000867. doi: 10.1136/bmjdrc-2019-000867. PMID 32475836
- See also: U.S. Census Bureau. (2013). 2013 American Community Survey 5-Year Estimates. — http://factfinder.census.gov/faces/tableservices/jsf/pages/productview.xhtml?pid=ACS_13_5YR_S0501&prodType=table